CLINICAL TRIAL: NCT01905709
Title: Fecal Microbiota Transplantation for the Treatment of Recurrent or Refractory Clostridium Difficile Infection (CDI)
Brief Title: Fecal Microbiota Transplantation for C Diff Infection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Englewood Hospital and Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E-13-507
Record Dates: First submitted 2013-07-19; First posted 2013-07-23 (Estimated); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Clostridium Difficile Infection
Keywords: C diff; CDI; clostridium difficile associated diarrhea
MeSH Terms: conditions — Clostridium Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- All patients (Experimental): 150-500 ml of human fecal matter
  Interventions: Biological: Human fecal matter

INTERVENTIONS:
Biological: Human fecal matter
  Other Names: human stool

SUMMARY:
The objective of this study is to provide treatment with Fecal Microbiota Transplantation (FMT) to patients with recurrent or refractory Clostridium difficile infection (CDI). It has been shown that good bacteria (like that found in the stool from a healthy donor) attack Clostridium difficile in multiple ways: they make substances that kill Clostridium difficile - and they attach to the surface of the colon lining, which prevents the Clostridium difficile toxin (poison) from attaching.

FMT involves infusing a mixture of saline and stool from a healthy donor into the bowel of the patient with CDI during a colonoscopy.

The method used to deliver the FMT will depend on individual characteristics of the subject and is at the discretion of the treating physician. FMT may be administered by the following methods.

* Colonoscopy: This method allows full endoscopic examination of the colon and exclusion of comorbid conditions (such as IBD, malignancy or microscopic colitis) which may have an impact on subject's treatment or response to therapy.
* Sigmoidoscopy: This method still allows infusion of the stool into a more proximal segment of the colon than an enema, but may not require sedation. This method may be beneficial in subjects who are elderly or multiparous and who may have difficulty retaining the material when given as enema. Sigmoidoscopic administration eliminates the additional risks associated with colonoscopy in subjects who may not have a clear indication for colonoscopy.
* Retention enema: This method may be preferable in younger subjects who have already had recent endoscopic evaluation, in subjects who prefer not to undergo endoscopy or in subjects with significant co morbidities and may not tolerate endoscopy.

The physician will administer 300-500 mL of the fecal suspension in aliquots of 60 mL, through the colonoscope or sigmoidoscope or 150 mL via retention enema. In cases of colonoscopic delivery, the material will be delivered to the most proximal point of insertion.

The subject is encouraged to retain stool for as long as possible.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 years old.
2. Subject has recurrent or relapsing CDI defined as:

   * At least three episodes of mild-to-moderate CDI and failure of a 6-8 week taper with vancomycin with or without an alternative antibiotic (e.g., rifaximin, nitazoxanide, fidaxomicin). OR
   * At least two episodes of severe CDI resulting in hospitalization and associated with significant morbidity. OR
   * Moderate CDI not responding to standard therapy (vancomycin) for at least a week. OR
   * Severe C. difficile infection with toxic megacolon, not responding to standard therapy or the use of IVIg.
3. Subject is willing and able to provide informed consent.
4. If a female of childbearing potential, subject has agreed to use an acceptable form of birth control for up to 4 weeks after FMT treatment.

Exclusion Criteria:

1. Subject is pregnant.
2. Subject is unable to comply with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-07; Primary Completion 2026-07 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
CDI recurrence | 8 weeks
  Number of patients who did/did not experience relapse in the 8 weeks post FMT

CONTACTS AND LOCATIONS:
Overall Officials: Marc Fiorillo, MD, Principal Investigator — Englewood Hospital and Medical Center
Locations (1):
- Englewood Hospital and Medical Center, Englewood, New Jersey, United States